CLINICAL TRIAL: NCT01270451
Title: Guidance in Diet and Physical Activity for Prevention of Weight Gain After Gastric Bypass Surgery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other); Norwegian Foundation for Health and Rehabilitation (Other)
Responsible Party: Principal Investigator, Oslo University Hospital, Anne-Marie Aas, Oslo University Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 08/302d, 2008/6365 (REK); 08/7772 (Other: Biobankregisteret); NCT01592591 (obsolete NCT alias)
Record Dates: First submitted 2011-01-04; First posted 2011-01-05 (Estimated); Last update posted 2014-10-23 (Estimated); Status verified 2014-10

CONDITIONS: Obesity
Keywords: Weight maintenance; Group counseling; Prevention of diseases
MeSH Terms: conditions — Obesity | interventions — Body Weight Maintenance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lifestyle group counseling (Other): Included patients will be randomised into two groups: to the intervention group or to the control group.
  Interventions: Other: Lifestyle intervention to prevent weight regain

INTERVENTIONS:
Other: Lifestyle intervention to prevent weight regain — To study if subjects receiving extra guidance in diet and physical activity experience less weight gain compared to a control group.
  Other Names: Weight maintenance; Prevention of insulin resistance; Prevention of diabetes; Prevention of cardiovascular disease

SUMMARY:
Primary Outcomes:

1. To study cross-sectional associations between diet, physical activity, T2DM and weight in subjects 2 yrs after surgery.
2. To study if subjects receiving extra guidance in diet and physical activity experience less weight gain compared to a control group.

   Secondary Outcomes:
3. To study the association between vit.D levels and T2DM.
4. To study the association between weight change and QOL.
5. To validate the new guidance strategy by recording food intake, energy expenditure and physical activity level.
6. To study if subjects receiving extra guidance in diet and physical activity experience other health effects compared to a control group.
7. To search for biomarkers that can identify people at risk of increasing weight post surgery

DETAILED DESCRIPTION:
Expected weight loss after GBP is 60-80% of the overweight. GBP is effective therapy against the obesity-related disorders, including T2DM. Some subjects start gaining weight within 12-18 months after surgery. Weight gain may again increase the risk for developing obesity-related disorders. Previous studies have found a link between vitamin D deficiencies and T2DM. Vitamin D levels will be monitored during the intervention. Studies have shown that patients who underwent GBP experienced a dramatic improvement in quality of life(QOL). After reaching maximum weight loss, many will slowly gain weight. For some people that means a decrease in QOL. In order to prevent weight gain it may be useful to provide additional follow-ups. Participants are randomised into two groups: Group A will receive extra guidance and follow-up, while Group B will continue with the existing scheme. Participants in Group A will over the next 2 yrs take part in frequent meetings. To assess dietary habits, physical activity patterns and QOL, food diaries, physical activity questionnaires and QOL questionnaires are used. Anthropometric and blood pressure measurements will be taken and blood samples will be collected at regular time intervals before and during the study. The results will be used to validate the effect of extra guidance, and to decide if this treatment shall be offered to all of our patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing gastric bypass surgery at OUH in the period January 2006 to June 2009 (recruited 24 ± 9 months following surgery)
* Willingness to participate at regular meetings at OUH

Exclusion Criteria:

* Patients who have experienced serious complications due to the bariatric surgery
* Patients who do not understand Norwegian
* Immobile patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2008-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Weight regain | 2 and 4 years postsurgery

SECONDARY OUTCOMES:
Changes in QOL, insulin resistance, diabetes, cardiovascular risk factors, nutritional status. | 2 and 4 years postsurgery

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Marie Aas, Phd, Principal Investigator — Department of Nutrition & Dietetics, Oslo University Hospital, Aker; Helga Refsum, Prof.,MD,PhD, Study Director — Dept. of Nutrition, University of Oslo (UiO)
Locations (1):
- Oslo University Hospital, Oslo, Oslo County, Norway

REFERENCES:
- [Derived] Hanvold SE, Vinknes KJ, Loken EB, Hjartaker A, Klungsoyr O, Birkeland E, Risstad H, Gulseth HL, Refsum H, Aas AM. Does Lifestyle Intervention After Gastric Bypass Surgery Prevent Weight Regain? A Randomized Clinical Trial. Obes Surg. 2019 Nov;29(11):3419-3431. doi: 10.1007/s11695-019-04109-7. PMID 31363961